CLINICAL TRIAL: NCT02784795
Title: A Phase 1b Study of LY3039478 in Combination With Other Anticancer Agents in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study of LY3039478 in Participants With Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to business considerations
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16209; I6F-MC-JJCD (Other: Eli Lilly and Company); 2015-004421-14 (EudraCT Number)
Record Dates: First submitted 2016-05-25; First posted 2016-05-27 (Estimated); Results first posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumor; Breast Cancer; Colon Cancer; Cholangiocarcinoma; Soft Tissue Sarcoma
Keywords: Notch Inhibitor
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Cholangiocarcinoma; Sarcoma | interventions — crenigacestat; LY2940680; abemaciclib; Cisplatin; Gemcitabine; Carboplatin; LY3023414

STUDY DESIGN:
Intervention Model Description: As per the study protocol design description, the study was conducted as multicenter, nonrandomized, open-label, Phase 1b study consisting of 5 separate, parallel dose escalations in patients with advanced/metastatic cancer from a variety of solid tumors followed by a dose-confirmation phase in specified tumor types.
Oversight: Data Monitoring Committee: No

ARMS (12):
- Part A: 25 milligram (mg) LY3039478 + 200 mg Taladegib (Cohort 1) (Experimental): 25 mg LY3039478 given orally 3 times per week (TIW) in combination with 200 mg taladegib given orally once daily (QD) on a 28 day cycle. A single dose of 200 mg taladegib was also be given on day 1 during a 3-day lead-in period for pharmacokinetic (PK) evaluation.
  Participants receiving benefit may continue until disease progression.
  Interventions: Drug: LY3039478; Drug: Taladegib
- Part B: 25 mg LY3039478 + 150 mg LY3023414 (Cohort 1 - Dose Escalation) (Experimental): 25 mg LY3039478 given orally TIW in combination with 150 mg LY3023414 given orally twice daily (BID) on a 28 day cycle. A single dose of 150 mg LY3023414 was also be given on day 1 during a 3-day lead-in period for PK evaluation.
  Participants receiving benefit may continue until disease progression.
  Interventions: Drug: LY3039478; Drug: LY3023414
- Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2) (Experimental): 50 mg LY3039478 given orally TIW in combination with 150 mg LY3023414 given orally twice daily (BID) on a 28 day cycle. A single dose of 150 mg LY3023414 was also be given on day 1 during a 3-day lead-in period for PK evaluation.
  Participants receiving benefit may continue until disease progression.
  Interventions: Drug: LY3039478; Drug: LY3023414
- Part B: 25 mg LY3039478 + 200 mg LY3023414 (Cohort 3) (Experimental): 25 mg LY3039478 given orally TIW in combination with 200 mg LY3023414 given orally twice daily (BID) on a 28 day cycle. A single dose of 200 mg LY3023414 was also be given on day 1 during a 3-day lead-in period for PK evaluation.
  Participants receiving benefit may continue until disease progression.
  Interventions: Drug: LY3039478; Drug: LY3023414
- Part B: 25 mg LY3039478 + 150 mg LY3023414 (Cohort 4 - Dose Confirmation) (Experimental): 25 mg LY3039478 given orally TIW in combination with 150 mg LY3023414 given orally twice daily (BID) on a 28 day cycle. A single dose of 150 mg LY3023414 was also be given on day 1 during a 3-day lead-in period for PK evaluation.
  Participants receiving benefit may continue until disease progression.
  Interventions: Drug: LY3039478; Drug: LY3023414
- Part C: 25 mg LY3039478 + 100 mg Abemaciclib (Cohort 1) (Experimental): 25 mg LY3039478 given orally TIW in combination with 100 mg abemaciclib given orally BID on a 28-day cycle. A single dose of 100 mg abemaciclib was also be given on day 1 during a 3-day lead-in period for PK evaluation.
  Participants receiving benefit may continue until disease progression.
  Interventions: Drug: LY3039478; Drug: Abemaciclib
- Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2) (Experimental): 50 mg LY3039478 given orally TIW in combination with 100 mg abemaciclib given orally BID on a 28-day cycle. A single dose of 100 mg abemaciclib was also be given on day 1 during a 3-day lead-in period for PK evaluation.
  Participants receiving benefit may continue until disease progression.
  Interventions: Drug: LY3039478; Drug: Abemaciclib
- Part C: 25 mg LY3039478 + 150 mg Abemaciclib (Cohort 3) (Experimental): 25 mg LY3039478 given orally TIW in combination with 150 mg abemaciclib given orally BID on a 28-day cycle. A single dose of 150 mg abemaciclib was also be given on day 1 during a 3-day lead-in period for PK evaluation.
  Participants receiving benefit may continue until disease progression.
  Interventions: Drug: LY3039478; Drug: Abemaciclib
- Part D:25 mg LY3039478+25 Milligram/Square Meter (mg/m2) Cisplatin+1000 mg/m2 Gemcitabine (Cohort 1) (Experimental): 25 mg LY3039478 given orally TIW in combination with 25 mg/m2 cisplatin and 1000 mg/m2 gemcitabine given as intravenous (IV) infusions on days 1 and 8 of a 21 day cycle.
  Participants receiving benefit may continue until disease progression.
  Interventions: Drug: LY3039478; Drug: Cisplatin; Drug: Gemcitabine
- Part D: 50 mg LY3039478 + 25 mg/m2 Cisplatin + 1000 mg/m2 Gemcitabine (Cohort 2) (Experimental): 50 mg LY3039478 given orally TIW in combination with 25 mg/m2 cisplatin and1000 mg/m2 gemcitabine given as IV infusions on days 1 and 8 of a 21 day cycle.
  Participants receiving benefit may continue until disease progression.
  Interventions: Drug: LY3039478; Drug: Cisplatin; Drug: Gemcitabine
- Part E: 25 mg LY3039478 + 1000 mg/m2 Gemcitabine + Carboplatin (Cohort 1) (Experimental): 25 mg LY3039478 given orally TIW in combination with 1000 mg/m2 gemcitabine and area under the plasma concentration-time curve dose of (AUC) carboplatin given as IV infusions on days 1 and 8 of a 21 day cycle.
  Participants receiving benefit may continue until disease progression.
  Interventions: Drug: LY3039478; Drug: Gemcitabine; Drug: Carboplatin
- Part E: 50 mg LY3039478 + 1000 mg/m2 Gemcitabine + Carboplatin (Cohort 2) (Experimental): 50 mg LY3039478 given orally TIW in combination with 1000 mg/m2 gemcitabine and AUC dose of carboplatin given as IV infusions on days 1 and 8 of a 21 day cycle.
  Participants receiving benefit may continue until disease progression.
  Interventions: Drug: LY3039478; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: LY3039478 — Administered orally
Drug: Taladegib — Administered orally
  Other Names: LY2940680
  Arms: Part A: 25 milligram (mg) LY3039478 + 200 mg Taladegib (Cohort 1)
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Part C: 25 mg LY3039478 + 100 mg Abemaciclib (Cohort 1); Part C: 25 mg LY3039478 + 150 mg Abemaciclib (Cohort 3); Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2)
Drug: Cisplatin — Administered IV
  Arms: Part D: 50 mg LY3039478 + 25 mg/m2 Cisplatin + 1000 mg/m2 Gemcitabine (Cohort 2); Part D:25 mg LY3039478+25 Milligram/Square Meter (mg/m2) Cisplatin+1000 mg/m2 Gemcitabine (Cohort 1)
Drug: Gemcitabine — Administered IV
  Arms: Part D: 50 mg LY3039478 + 25 mg/m2 Cisplatin + 1000 mg/m2 Gemcitabine (Cohort 2); Part D:25 mg LY3039478+25 Milligram/Square Meter (mg/m2) Cisplatin+1000 mg/m2 Gemcitabine (Cohort 1); Part E: 25 mg LY3039478 + 1000 mg/m2 Gemcitabine + Carboplatin (Cohort 1); Part E: 50 mg LY3039478 + 1000 mg/m2 Gemcitabine + Carboplatin (Cohort 2)
Drug: Carboplatin — Administered IV
  Arms: Part E: 25 mg LY3039478 + 1000 mg/m2 Gemcitabine + Carboplatin (Cohort 1); Part E: 50 mg LY3039478 + 1000 mg/m2 Gemcitabine + Carboplatin (Cohort 2)
Drug: LY3023414 — Administered orally
  Arms: Part B: 25 mg LY3039478 + 150 mg LY3023414 (Cohort 1 - Dose Escalation); Part B: 25 mg LY3039478 + 150 mg LY3023414 (Cohort 4 - Dose Confirmation); Part B: 25 mg LY3039478 + 200 mg LY3023414 (Cohort 3); Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2)

SUMMARY:
The main purpose of this study is to evaluate the safety of the study drug known as LY3039478 in combination with other anticancer agents in participants with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* For all parts: The participant must be, in the judgment of the investigator, an appropriate candidate for experimental therapy after available standard therapies have failed to provide clinical benefit for their advanced or metastatic cancer.

  * For dose escalation for all combinations: The participant must have histological or cytological evidence of cancer, either a solid tumor or a lymphoma, which is advanced or metastatic.
  * For Part A dose confirmation: All participants must have histological evidence of advanced or metastatic soft tissue sarcoma or breast cancer. Breast cancer participants must have prescreened mutations, amplification, or gene/protein expression alterations related to Notch pathway.
  * For Part B dose confirmation: All participants must have histological evidence of advanced or metastatic colon cancer or soft tissue sarcoma. Colon cancer participants must have prescreened mutations, amplification, or gene/protein expression alterations related to Notch pathway.
  * For Part C dose confirmation: All participants must have histological evidence of advanced or metastatic breast cancer and prescreened mutations, amplification, or gene/protein expression alterations related to Notch pathway.
  * For Part D dose confirmation: All participants must have histological evidence of cholangiocarcinoma and prescreened mutations, amplification, or gene/protein expression alterations related to Notch pathway. Participants must not have received >1 line of prior systemic therapy for metastatic or resectable disease (that is, participants may have received adjuvant gemcitabine and then later gemcitabine/cisplatin for recurrent metastatic disease).
  * For Part E dose confirmation: All participants must have histological evidence of locally advanced or metastatic triple negative breast cancer (TNBC) and prescreened mutations, amplification, or gene/protein expression alterations related to Notch pathway. Participants must not have received >2 lines of systemic treatment for advanced or metastatic TNBC.
* Have adequate organ function.
* Have a performance status of ≤1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have discontinued all previous therapies for cancer.

Exclusion Criteria:

* Have current acute leukemia.
* Have current or recent (within 3 months of study drug administration) gastrointestinal disease with chronic or intermittent diarrhea, or disorders that increase the risk of diarrhea, such as inflammatory bowel disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- United States (4):
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Rigshospitalet, Copenhagen, København Ø, Denmark
- France (3):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Gustave Roussy, Villejuif
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid

REFERENCES:
- [Derived] Massard C, Cassier PA, Azaro A, Anderson B, Yuen E, Yu D, Oakley G 3rd, Benhadji KA, Pant S. A phase 1b study of crenigacestat (LY3039478) in combination with gemcitabine and cisplatin or gemcitabine and carboplatin in patients with advanced or metastatic solid tumors. Cancer Chemother Pharmacol. 2022 Oct;90(4):335-344. doi: 10.1007/s00280-022-04461-z. Epub 2022 Aug 28. PMID 36030462
- [Derived] Azaro A, Massard C, Tap WD, Cassier PA, Merchan J, Italiano A, Anderson B, Yuen E, Yu D, Oakley G 3rd, Benhadji KA, Pant S. A phase 1b study of the Notch inhibitor crenigacestat (LY3039478) in combination with other anticancer target agents (taladegib, LY3023414, or abemaciclib) in patients with advanced or metastatic solid tumors. Invest New Drugs. 2021 Aug;39(4):1089-1098. doi: 10.1007/s10637-021-01094-6. Epub 2021 Mar 8. PMID 33686452
- See also: Click here for more information about this study:A Study of LY3039478 in Participants With Advanced or Metastatic Solid Tumors — https://lillytrialguide.com/en/studies/solid-tumor/JJCD#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consists of 5 separate, parallel dose escalations (dose esc) followed by dose-confirmation (dose conf) study parts (Part A - E). LY3039478 is given in combination with taladegib for Part A, LY3023414 for Part B, abemaciclib (abema) for Part C, cisplatin (cis) and gemcitabine (gem) for Part C, and gemcitabine and carboplatin (carb) for Part E. A participant completed the study if they completed at least 1 cycle (1 cycle = 28 days for Part A, B and C and 21 days for Part D, E) .
Groups:
- Part A:25 Milligram(mg) LY3039478+200 mg Taladegib(Cohort 1): 25 mg LY3039478 given orally 3 times per week (TIW) in combination with 200 mg taladegib given orally once daily (QD) on a 28 day cycle. A single dose of 200 mg taladegib was also be given on day 1 during a 3-day lead-in period for pharmacokinetic (PK) evaluation.
  Participants receiving benefit may continue until disease progression.
- Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 1-Dose Esc); Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 4-Dose Conf): 25 mg LY3039478 given orally TIW in combination with 150 mg LY3023414 given orally twice daily (BID) on a 28 day cycle. A single dose of 150 mg LY3023414 was also be given on day 1 during a 3-day lead-in period for PK evaluation.
  Participants receiving benefit may continue until disease progression.
- Part D:25 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem (Cohort 1): 25 mg LY3039478 given orally TIW in combination with 25 mg/m2 cisplatin and 1000 mg/m2 gemcitabine given as intravenous (IV) infusions on days 1 and 8 of a 21 day cycle.
  Participants receiving benefit may continue until disease progression.
- Part D:50 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem(Cohort 2): 50 mg LY3039478 given orally TIW in combination with 25 mg/m2 cisplatin and1000 mg/m2 gemcitabine given as IV infusions on days 1 and 8 of a 21 day cycle.
  Participants receiving benefit may continue until disease progression
- Part E:25 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 1): 25 mg LY3039478 given orally TIW in combination with 1000 mg/m2 gemcitabine and area under the plasma concentration-time curve dose of (AUC) carboplatin given as IV infusions on days 1 and 8 of a 21 day cycle.
  Participants receiving benefit may continue until disease progression.
- Part E:50 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 2): 50 mg LY3039478 given orally TIW in combination with 1000 mg/m2 gemcitabine and AUC dose of carboplatin given as IV infusions on days 1 and 8 of a 21 day cycle.
  Participants receiving benefit may continue until disease progression.
Period: Overall Study
Arm/Group | Part A:25 Milligram(mg) LY3039478+200 mg Taladegib(Cohort 1) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 1-Dose Esc) | Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2) | Part B: 25 mg LY3039478 + 200 mg LY3023414 (Cohort 3) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 4-Dose Conf) | Part C: 25 mg LY3039478 + 100 mg Abemaciclib (Cohort 1) | Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2) | Part C: 25 mg LY3039478 + 150 mg Abemaciclib (Cohort 3) | Part D:25 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem (Cohort 1) | Part D:50 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem(Cohort 2) | Part E:25 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 1) | Part E:50 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 2)
Started | 8 | 5 | 4 | 5 | 18 | 3 | 12 | 8 | 6 | 10 | 5 | 10
Received at Least One Dose of Study Drug | 8 | 5 | 4 | 5 | 18 | 3 | 12 | 8 | 6 | 10 | 5 | 10
Completed at Least 1 Treatment Cycle | 8 | 5 | 4 | 5 | 18 | 3 | 12 | 8 | 6 | 10 | 5 | 10
Completed | 4 | 4 | 1 | 3 | 12 | 3 | 8 | 7 | 6 | 10 | 4 | 6
Not Completed | 4 | 1 | 3 | 2 | 6 | 0 | 4 | 1 | 0 | 0 | 1 | 4
Not completed — Progressive Disease | 2 | 1 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants in Part A, B, C, D and E.
Groups:
- Part A:25 mg LY3039478+200 mg Taladegib(Cohort 1): 25 mg LY3039478 given orally TIW in combination with 200 mg taladegib given orally QD on a 28 day cycle.
  Participants receiving benefit may continue until disease progression.
- Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 1-Dose Esc); Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 4-Dose Conf): 25 mg LY3039478 given orally TIW in combination with 150 mg LY3023414 given orally BID on a 28 day cycle.
  Participants receiving benefit may continue until disease progression.
- Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2): 50 mg LY3039478 given orally TIW in combination with 150 mg LY3023414 given orally BID on a 28 day cycle.
  Participants receiving benefit may continue until disease progression.
- Part B: 25 mg LY3039478 + 200 mg LY3023414 (Cohort 3): 25 mg LY3039478 given orally TIW in combination with 200 mg LY3023414 given orally BID on a 28 day cycle.
  Participants receiving benefit may continue until disease progression.
- Part C: 25 mg LY3039478 + 100 mg Abemaciclib (Cohort 1): 25 mg LY3039478 given orally TIW in combination with 100 mg abemaciclib given orally BID on a 28-day cycle.
  Participants receiving benefit may continue until disease progression.
- Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2): 50 mg LY3039478 given orally TIW in combination with 100 mg abemaciclib given orally BID on a 28-day cycle.
  Participants receiving benefit may continue until disease progression.
- Part C: 25 mg LY3039478 + 150 mg Abemaciclib (Cohort 3): 25 mg LY3039478 given orally TIW in combination with 150 mg abemaciclib given orally BID on a 28-day cycle.
  Participants receiving benefit may continue until disease progression.
- Total: Total of all reporting groups
Arm/Group | Part A:25 mg LY3039478+200 mg Taladegib(Cohort 1) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 1-Dose Esc) | Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2) | Part B: 25 mg LY3039478 + 200 mg LY3023414 (Cohort 3) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 4-Dose Conf) | Part C: 25 mg LY3039478 + 100 mg Abemaciclib (Cohort 1) | Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2) | Part C: 25 mg LY3039478 + 150 mg Abemaciclib (Cohort 3) | Part D:25 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem (Cohort 1) | Part D:50 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem(Cohort 2) | Part E:25 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 1) | Part E:50 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 2) | Total
Number analyzed (Participants) | 8 | 5 | 4 | 5 | 18 | 3 | 12 | 8 | 6 | 10 | 5 | 10 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (16.8) | 53.0 (8.5) | 62.3 (3.9) | 56.6 (11.8) | 47.2 (13.4) | 60.0 (11.8) | 54.3 (11.4) | 51.1 (13.9) | 59.7 (8.6) | 52.6 (12.9) | 62.8 (6.8) | 53.6 (12.2) | 54.0 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 3 | 12 | 2 | 8 | 4 | 3 | 5 | 4 | 8 | 54
  Male | 6 | 3 | 3 | 2 | 6 | 1 | 4 | 4 | 3 | 5 | 1 | 2 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 4 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 10
  Not Hispanic or Latino | 7 | 5 | 3 | 5 | 13 | 3 | 11 | 5 | 5 | 9 | 5 | 7 | 78
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  White | 7 | 4 | 3 | 5 | 13 | 3 | 11 | 6 | 6 | 9 | 5 | 6 | 78
  More than one race | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 2 | 2 | 9 | 0 | 7 | 0 | 1 | 3 | 0 | 4 | 34
  Denmark | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  France | 3 | 0 | 2 | 2 | 4 | 1 | 3 | 4 | 3 | 6 | 3 | 5 | 36
  Spain | 2 | 2 | 0 | 1 | 4 | 2 | 2 | 4 | 2 | 1 | 2 | 1 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With LY3039478 Dose-Limiting Toxicities (DLT) in Part A, B, C, D and E
Description: DLT is defined as an adverse event (AE) during Cycle 1 (28 days for Part A, B and C and 21 days for Part D, E) that was possibly related to the study drug and met 1 of the following criteria: According to the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0: ≥Grade 3 non-hematological toxicity except nausea/vomiting, diarrhea, or constipation that can be controlled with appropriate care; Grade 3 elevations of alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) lasting fewer than 8 days (without evidence of other hepatic injury); Grade 3 rash that resolves or improves to a Grade 2 or less within 7 days; CTCAE Grade 4 hematological toxicity of >5 days duration; Grade 4 thrombocytopenia of any duration; Grade 3 thrombocytopenia with bleeding; Grade 3 febrile neutropenia.
Time Frame: Baseline to toxicity (up to end of Cycle 1 [1Cycle = 28 days for Part A, B and C and 21 days for Part D, E])
Population: All participants who receive at least one dose of study drug in Part A, B, C, D and E.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A:25 mg LY3039478+200 mg Taladegib(Cohort 1) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 1-Dose Esc) | Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2) | Part B: 25 mg LY3039478 + 200 mg LY3023414 (Cohort 3) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 4-Dose Conf) | Part C: 25 mg LY3039478 + 100 mg Abemaciclib (Cohort 1) | Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2) | Part C: 25 mg LY3039478 + 150 mg Abemaciclib (Cohort 3) | Part D:25 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem (Cohort 1) | Part D:50 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem(Cohort 2) | Part E:25 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 1) | Part E:50 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 2)
Number analyzed (Participants) | 8 | 5 | 4 | 5 | 18 | 3 | 12 | 8 | 6 | 10 | 5 | 10
Participants | 2 | 0 | 2 | 3 | 3 | 0 | 2 | 0 | 1 | 3 | 2 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC[0-∞]) of LY3039478 in Combination With Taladegib, LY3023414, Abemaciclib, Cisplatin/Gemcitabine, and Gemcitabine/Carboplatin in Part A, B, C, D and E
Description: AUC[0-∞] of LY3039478 in combination with taladegib, LY3023414, abemaciclib, cisplatin/gemcitabine, and gemcitabine/carboplatin in dose escalation parts of Part A, B, C, D and E was evaluated.
Time Frame: Parts A/B/C Day 22 (Cycle 1): pre-dose, 0.5, 1, 2, 4, 6, 8, 24-30 hours post-dose; Parts D/E Day 1 (Cycle 1) and 15 (Cycle 1): pre-dose, 0.5, 1, 2, 4, 6-8, 24-30 hours post-dose
Population: All participants who received at least one dose of study drug with intensive PK sampling in the dose escalation cohorts of Part A, B, C, D and E. PK data was interpreted by combining Part B (25 mg LY3039478 + 150/200 mg LY3023414; Cohorts 1 and 3) and Part C (25 mg LY3039478 + 100/150 mg abemaciclib; Cohorts 1 and 3) reporting arms as all participants received same dose of 50 mg LY3039478 (Part B and C Cohorts 1 and 2) and to increase the sample size for interpretability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/mL (ng*h/mL)
Groups:
- Part A:25 mg LY3039478+200 mg Taladegib(Cohort 1): 25 mg LY3039478 given orally TIW in combination with 200 mg taladegib given orally QD on a 28 day cycle. A single dose of 200 mg taladegib was also be given on day 1 during a 3-day lead-in period.
  Participants receiving benefit may continue until disease progression.
- Part B:25 mg LY3039478+150mg/200 mg LY3023414(Cohort 1 and 3): 25 mg LY3039478 given orally TIW in combination with 150 mg LY3023414 given orally BID on a 28 day cycle. A single dose of 150 mg LY3023414 was also be given on day 1 during a 3-day lead-in period in cohort 1 and 25 mg LY3039478 given orally TIW in combination with 200 mg LY3023414 given orally BID on a 28 day cycle in cohort 3.
  Participants receiving benefit may continue until disease progression.
- Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2): 50 mg LY3039478 given orally TIW in combination with 150 mg LY3023414 given orally BID on a 28 day cycle. A single dose of 150 mg LY3023414 was also be given on day 1 during a 3-day lead-in period.
  Participants receiving benefit may continue until disease progression.
- Part C:25 mg LY3039478+100 mg/150 mg Abema(Cohort 1 and 3): 25 mg LY3039478 given orally TIW in combination with 100 mg abemaciclib given orally BID on a 28-day cycle. A single dose of 100 mg abemaciclib was also be given on day 1 during a 3-day lead-in period in cohort 1 and 25 mg LY3039478 given orally TIW in combination with 150 mg abemaciclib given orally BID on a 28-day cycle in cohort 3.
  Participants receiving benefit may continue until disease progression.
- Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2): 50 mg LY3039478 given orally TIW in combination with 100 mg abemaciclib given orally BID on a 28-day cycle. A single dose of 100 mg abemaciclib was also be given on day 1 during a 3-day lead-in period.
  Participants receiving benefit may continue until disease progression.
Arm/Group | Part A:25 mg LY3039478+200 mg Taladegib(Cohort 1) | Part B:25 mg LY3039478+150mg/200 mg LY3023414(Cohort 1 and 3) | Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2) | Part C:25 mg LY3039478+100 mg/150 mg Abema(Cohort 1 and 3) | Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2) | Part D:25 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem (Cohort 1) | Part D:50 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem(Cohort 2) | Part E:25 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 1) | Part E:50 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 2)
Number analyzed (Participants) | 1 | 6 | 1 | 4 | 4 | 4 | 7 | 2 | 7
nanogram*hour/mL (ng*h/mL)
  Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 4 | 7 | 1 | 7
  Day 1 |  |  |  |  |  | 1210 (41) | 3080 (35) | NA (NA) — AUC[0-∞] could not be calculated for one participant in the "Part E:25 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 1)" Arm for the Day 1 | 3400 (70)
  Day 15: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 2
  Day 15 |  |  |  |  |  | 1030 (9) | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual value = 1980 ng*h/mL. | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual range = 804 -1400 ng*h/mL. | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual range = 3350 - 3620 ng*h/mL.
  Day 22: number analyzed (Participants) | 1 | 6 | 1 | 4 | 4 | 0 | 0 | 0 | 0
  Day 22 | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual value = 295 ng*h/mL. | 2660 (31) | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual value = 4250 ng*h/mL. | 1820 (44) | 5080 (12) |  |  |  |

3. Secondary Outcome: PK: AUC[0-∞] of Taladegib and Its Active Metabolite LSN3185556, in Combination With LY3039478 (Part A)
Description: AUC[0-∞] of taladegib and its active metabolite LSN3185556, in combination with LY3039478 (Part A) was evaluated.
Time Frame: Day -3 (Lead in) : pre-dose, 0.5, 1, 2, 4, 6, 8, 24-30, 72 hours post-dose and Day 22 (Cycle 1): pre-dose, 0.5, 1, 2, 4, 6, 8, 24 hours post-dose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A:25 mg LY3039478+200 mg Taladegib(Cohort 1)
Number analyzed (Participants) | 6
ng*h/mL
  Taladegib: Day -3 | 17100 (48)
  Taladegib: Day 22: number analyzed (Participants) | 1
  Taladegib: Day 22 | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual value = 15400 ng*h/mL.
  LSN3185556 (Metabolite): Day -3: number analyzed (Participants) | 3
  LSN3185556 (Metabolite): Day -3 | 31900 (49)
  LSN3185556 (Metabolite): Day 22: number analyzed (Participants) | 1
  LSN3185556 (Metabolite): Day 22 | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual value = 26400 ng*h/mL.

4. Secondary Outcome: PK: AUC[0-∞] of LY3023414 in Combination With LY3039478 on Day -3 (Part B)
Description: AUC[0-∞] of LY3023414 in combination with LY3039478 (Part B) on day -3 was evaluated.
Time Frame: Day -3 (Lead in): pre-dose, 0.5, 1, 2, 4, 6, 8, 24-30, 72 hours post-dose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data in Part B. Day -3 Cohort 1 and 2 results for Parts B were combined as 'Part B:150 mg LY3023414 (Cohort 1 and Cohort 2)' since they are from same dose and were collected in the absence of LY3039478 co-administration. Part B Cohort 4 participants had sparse PK sampling limited to day 22 so day -3 PK results are not available/reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Part B:150 mg LY3023414 (Cohort 1 and Cohort 2): A single dose of 150 mg LY3023414 was given on day 1 during a 3-day lead-in period.
- Part B: 200 mg LY3023414 (Cohort 3): A single dose of 200 mg LY3023414 was given on day 1 during a 3-day lead-in period.
  Participants receiving benefit may continue until disease progression.
Arm/Group | Part B:150 mg LY3023414 (Cohort 1 and Cohort 2) | Part B: 200 mg LY3023414 (Cohort 3)
Number analyzed (Participants) | 8 | 5
ng*h/mL | 2620 (52) | 2780 (69)

5. Secondary Outcome: PK: AUC[0-∞] of LY3023414 in Combination With LY3039478 on Day 22 (Part B)
Description: AUC[0-∞] of LY3023414 in combination with LY3039478 (Part B) on day 22 was evaluated. LY3023414 PK data is summarized only for dose escalation patients in Part B with intensive PK sampling.
Time Frame: Day 22 (Cycle 1): pre-dose, 0.5, 1, 2, 4, 6, 8 hours post-dose
Population: All participants who received at least one dose of study drug with intensive PK sampling in the dose escalation cohort of Part B
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 1-Dose Esc) | Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2) | Part B: 25 mg LY3039478 + 200 mg LY3023414 (Cohort 3)
Number analyzed (Participants) | 4 | 1 | 2
ng*h/mL | 2120 (50) | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual value = 2480 ng*h/mL. | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual range value = 2900 - 12000 ng*h/mL.

6. Secondary Outcome: PK: AUC[0-∞] of Abemaciclib and AUC From Time Zero to the Last Measured Concentration Value (AUC[0-tlast]) of Its Major Active Metabolites LSN2839567 and LSN3106726, in Combination With LY3039478 on Day -3 (Part C)
Description: AUC[0-∞] of abemaciclib and AUC[0-tlast] of its major active metabolites LSN2839567 and LSN3106726, in combination with LY3039478 on Day 3 (Part C) was evaluated.
Time Frame: Day -3 (Lead in): pre-dose, 0.5, 1, 2, 4, 6, 8, 24-30, 72 hours post-dose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data in Part C. Day -3 Cohort 1 and 2 results for Parts B were combined as Part C: 100 mg Abemaciclib (Cohort 1 and Cohort 2) since they are from same dose and were collected in the absence of LY3039478 co-administration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Part C:100 mg Abemaciclib (Cohort 1 and Cohort 2): A single dose of 100 mg abemaciclib was given on day 1 during a 3-day lead-in period.
- Part C:150 mg Abemaciclib (Cohort 3): A single dose of 150 mg abemaciclib was given on day 1 during a 3-day lead-in period.
  Participants receiving benefit may continue until disease progression.
Arm/Group | Part C:100 mg Abemaciclib (Cohort 1 and Cohort 2) | Part C:150 mg Abemaciclib (Cohort 3)
Number analyzed (Participants) | 13 | 6
ng*h/mL
  Abemaciclib: number analyzed (Participants) | 12 | 5
  Abemaciclib | 4570 (78) | 3240 (109)
  LSN2839567 (Metabolite) | 778 (65) | 663 (82)
  LSN3106726 (Metabolite) | 1700 (59) | 1510 (76)

7. Secondary Outcome: PK: AUC[0-∞] of Abemaciclib and AUC From Time Zero to the Last Measured Concentration Value (AUC[0-tlast]) of Its Major Active Metabolites LSN2839567 and LSN3106726, in Combination With LY3039478 on Day 22 (Part C)
Description: AUC[0-∞] of abemaciclib and AUC[0-tlast] of its major active metabolites LSN2839567 and LSN3106726, in combination with LY3039478 on Day 22 (Part C) was evaluated.
Time Frame: Day 22 (Cycle 1): pre-dose, 0.5, 1, 2, 4, 6, 8 hours post-dose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data in Part C.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part C: 25 mg LY3039478 + 100 mg Abemaciclib (Cohort 1) | Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2) | Part C: 25 mg LY3039478 + 150 mg Abemaciclib (Cohort 3)
Number analyzed (Participants) | 3 | 2 | 1
ng*h/mL
  Abemaciclib | 5270 (88) | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual range value = 2510 - 6370 ng*h/mL. | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual value = 3420 ng*h/mL.
  LSN2839567 (Metabolite): number analyzed (Participants) | 3 | 1 | 1
  LSN2839567 (Metabolite) | 1460 (82) | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual value = 2130 ng*h/mL. | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual value = 914 ng*h/mL.
  LSN3106726 (Metabolite): number analyzed (Participants) | 2 | 1 | 1
  LSN3106726 (Metabolite) | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual range value = 2150 - 2690 ng*h/mL. | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual value = 4120 ng*h/mL. | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual value = 2590 ng*h/mL.

8. Secondary Outcome: Duration of Response (DoR)
Description: DoR was the time from the date of first evidence of complete response or partial response to the date of objective progression or the date of death due to any cause, whichever is earlier. CR and PR were defined using the RECIST v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. If a responder was not known to have died or have objective progression as of the data inclusion cutoff date, duration of response was censored at the last adequate tumor assessment date.
Time Frame: Date of Complete Response (CR) or Partial Response (PR) to Date of Objective Disease Progression (Up To 12 Months)
Population: Duration of Response was not calculated for any participant as the study was terminated prior to data collection.
Arm/Group | Part A:25 mg LY3039478+200 mg Taladegib(Cohort 1) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 1-Dose Esc) | Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2) | Part B: 25 mg LY3039478 + 200 mg LY3023414 (Cohort 3) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 4-Dose Conf) | Part C: 25 mg LY3039478 + 100 mg Abemaciclib (Cohort 1) | Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2) | Part C: 25 mg LY3039478 + 150 mg Abemaciclib (Cohort 3) | Part D:25 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem (Cohort 1) | Part D:50 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem(Cohort 2) | Part E:25 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 1) | Part E:50 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 2)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Progression Free Survival (PFS) Time in Part A, B, C, D and E
Description: PFS defined as the time from the date of randomization to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of randomization, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date. PFS time was summarized using Kaplan-Meier estimates.
Time Frame: Baseline to Objective Disease Progression or Death (Up To 1.91 Months for Part A, 7.69 Months for Part B, 11.53 Months for Part C, 19.52 Months for Part D, 7.03 Months for Part E)
Population: All randomized participants in Part A, B, C, D and E. Censored participants: Part A= 2, Part B = 0, 4, 2 and 7, Part C = 0, 6 and 5, Part D = 2, 3, Part E = 3, 7.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A:25 mg LY3039478+200 mg Taladegib(Cohort 1) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 1-Dose Esc) | Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2) | Part B: 25 mg LY3039478 + 200 mg LY3023414 (Cohort 3) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 4-Dose Conf) | Part C: 25 mg LY3039478 + 100 mg Abemaciclib (Cohort 1) | Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2) | Part C: 25 mg LY3039478 + 150 mg Abemaciclib (Cohort 3) | Part D:25 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem (Cohort 1) | Part D:50 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem(Cohort 2) | Part E:25 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 1) | Part E:50 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 2)
Number analyzed (Participants) | 8 | 5 | 4 | 5 | 18 | 3 | 12 | 8 | 6 | 10 | 5 | 10
Months | 1.22 [0.59 to 1.91] | 1.91 [1.35 to 2.00] | NA [NA to NA] — There were no events in Part B of Cohort 2. | 1.91 [1.87 to 7.69] | 1.84 [0.92 to 3.68] | 1.94 [1.61 to 11.53] | 1.91 [1.38 to 5.72] | NA [1.74 to NA] — The upper limit of the 95% confidence Interval (CI) was not calculated due to the high censoring rate. | 3.22 [2.96 to NA] — The upper limit of the 95% confidence Interval (CI) was not calculated due to the high censoring rate. | 3.02 [1.15 to 3.48] | 6.00 [4.96 to 7.03] | 4.71 [3.06 to 6.21]

ADVERSE EVENTS:
Time Frame: Up To 2 Months for Part A, 8 Months for Part B, 12 Months for Part C, 39 Months for Part D and 10 Months for Part E
Description: All randomized participants who received at least one dose of study drug in Part A, B, C, D and E. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Part A:25 mg LY3039478+200 mg Taladegib(Cohort 1): 25 mg LY3039478 given orally 3 times per week (TIW) in combination with 200 mg taladegib given orally once daily (QD) on a 28 day cycle.
  Participants receiving benefit may continue until disease progression.
- Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 1-Dose Esc); Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 4-Dose Conf): 25 mg LY3039478 given orally TIW in combination with 150 mg LY3023414 given orally twice daily (BID) on a 28 day cycle.
  Participants receiving benefit may continue until disease progression.
- Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2): 50 mg LY3039478 given orally TIW in combination with 150 mg LY3023414 given orally twice daily (BID) on a 28 day cycle.
  Participants receiving benefit may continue until disease progression.
- Part B: 25 mg LY3039478 + 200 mg LY3023414 (Cohort 3): 25 mg LY3039478 given orally TIW in combination with 200 mg LY3023414 given orally twice daily (BID) on a 28 day cycle.
  Participants receiving benefit may continue until disease progression.
Arm/Group | Part A:25 mg LY3039478+200 mg Taladegib(Cohort 1) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 1-Dose Esc) | Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2) | Part B: 25 mg LY3039478 + 200 mg LY3023414 (Cohort 3) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 4-Dose Conf) | Part C: 25 mg LY3039478 + 100 mg Abemaciclib (Cohort 1) | Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2) | Part C: 25 mg LY3039478 + 150 mg Abemaciclib (Cohort 3) | Part D:25 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem (Cohort 1) | Part D:50 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem(Cohort 2) | Part E:25 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 1) | Part E:50 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 3/8 | 1/5 | 0/4 | 0/5 | 9/18 | 1/3 | 1/12 | 1/8 | 0/6 | 0/10 | 0/5 | 0/10
Serious Adverse Events (participants affected / at risk) | 5/8 | 2/5 | 2/4 | 2/5 | 9/18 | 2/3 | 9/12 | 2/8 | 2/6 | 5/10 | 2/5 | 7/10
Other Adverse Events (participants affected / at risk) | 7/8 | 5/5 | 4/4 | 5/5 | 17/18 | 3/3 | 11/12 | 8/8 | 6/6 | 10/10 | 5/5 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A:25 mg LY3039478+200 mg Taladegib(Cohort 1) (N=8) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 1-Dose Esc) (N=5) | Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2) (N=4) | Part B: 25 mg LY3039478 + 200 mg LY3023414 (Cohort 3) (N=5) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 4-Dose Conf) (N=18) | Part C: 25 mg LY3039478 + 100 mg Abemaciclib (Cohort 1) (N=3) | Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2) (N=12) | Part C: 25 mg LY3039478 + 150 mg Abemaciclib (Cohort 3) (N=8) | Part D:25 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem (Cohort 1) (N=6) | Part D:50 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem(Cohort 2) (N=10) | Part E:25 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 1) (N=5) | Part E:50 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 2) (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A:25 mg LY3039478+200 mg Taladegib(Cohort 1) (N=8) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 1-Dose Esc) (N=5) | Part B: 50 mg LY3039478 + 150 mg LY3023414 (Cohort 2) (N=4) | Part B: 25 mg LY3039478 + 200 mg LY3023414 (Cohort 3) (N=5) | Part B:25 mg LY3039478+150 mg LY3023414 (Cohort 4-Dose Conf) (N=18) | Part C: 25 mg LY3039478 + 100 mg Abemaciclib (Cohort 1) (N=3) | Part C: 50 mg LY3039478 + 100 mg Abemaciclib (Cohort 2) (N=12) | Part C: 25 mg LY3039478 + 150 mg Abemaciclib (Cohort 3) (N=8) | Part D:25 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem (Cohort 1) (N=6) | Part D:50 mg LY3039478+25 mg/m2 Cis+1000 mg/m2 Gem(Cohort 2) (N=10) | Part E:25 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 1) (N=5) | Part E:50 mg LY3039478 + 1000 mg/m2 Gem + Carb (Cohort 2) (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 3 (6) | 1 (1) | 2 (3) | 4 (5) | 3 (8) | 1 (1) | 5 (7) | 5 (21) | 6 (12) | 4 (23) | 6 (25)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 2 (6) | 3 (6) | 4 (16) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (6) | 2 (4) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelash discolouration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Xerophthalmia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 2 (6) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (5) | 4 (7) | 3 (5) | 1 (6) | 10 (16) | 3 (16) | 8 (13) | 6 (19) | 5 (20) | 7 (15) | 3 (13) | 9 (25)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (4) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (10) | 4 (6) | 2 (4) | 5 (8) | 15 (22) | 3 (4) | 7 (9) | 4 (13) | 6 (34) | 9 (20) | 4 (11) | 7 (30)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (8) | 7 (13) | 0 (0) | 1 (2) | 2 (2) | 2 (2) | 2 (3) | 2 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 4 (11) | 2 (3) | 4 (10) | 10 (15) | 2 (6) | 3 (3) | 7 (9) | 5 (14) | 7 (18) | 4 (7) | 4 (19)
Asthenia (General disorders) | 3 (4) | 1 (3) | 0 (0) | 1 (1) | 3 (4) | 2 (3) | 1 (1) | 3 (8) | 2 (5) | 3 (4) | 2 (6) | 1 (1)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1) | 2 (3) | 3 (3) | 4 (7) | 1 (2) | 4 (8) | 4 (7) | 4 (14) | 5 (13) | 2 (3) | 2 (5)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 2 (2)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bartholin's abscess (Infections and infestations) | 0/2 (0) | 0/2 (0) | 0/1 (0) | 0/3 (0) | 0/12 (0) | 0/2 (0) | 0/8 (0) | 0/4 (0) | 0/3 (0) | 1/5 (1) | 0/4 (0) | 0/8 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0/2 (0) | 0/2 (0) | 0/1 (0) | 0/3 (0) | 1/12 (1) | 0/2 (0) | 0/8 (0) | 0/4 (0) | 0/3 (0) | 0/5 (0) | 0/4 (0) | 0/8 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0/2 (0) | 0/2 (0) | 0/1 (0) | 0/3 (0) | 0/12 (0) | 0/2 (0) | 0/8 (0) | 0/4 (0) | 0/3 (0) | 0/5 (0) | 0/4 (0) | 1/8 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 2 (7) | 5 (11) | 2 (3) | 3 (6) | 1 (1) | 4 (8) | 5 (12) | 4 (13) | 5 (13)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 2 (7) | 4 (8) | 3 (4) | 3 (6) | 1 (1) | 3 (5) | 4 (8) | 4 (7) | 6 (13)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (4) | 1 (1) | 5 (9) | 1 (1) | 2 (5) | 1 (1) | 0 (0)
Blood culture positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 1 (3) | 1 (1) | 0 (0) | 2 (7) | 1 (1) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (2) | 1 (2) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (19) | 1 (1) | 2 (6) | 1 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (13) | 4 (11) | 4 (15) | 4 (15)
Nutritional condition abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (31) | 7 (25) | 3 (14) | 5 (30)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 2 (10) | 2 (3) | 0 (0) | 2 (3)
Weight increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (15) | 2 (4) | 0 (0) | 2 (6)
Appetite disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 2 (2) | 3 (8) | 6 (7) | 2 (2) | 3 (3) | 5 (10) | 4 (12) | 3 (6) | 1 (1) | 3 (13)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (2) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (10) | 0 (0) | 0 (0) | 1 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (6) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (5) | 1 (6) | 1 (1) | 6 (14) | 2 (3) | 3 (6) | 3 (7) | 2 (3) | 2 (3) | 0 (0) | 4 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 4 (5) | 2 (3) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 3 (10) | 2 (5) | 2 (8) | 11 (14) | 3 (7) | 4 (17) | 5 (11) | 5 (47) | 7 (21) | 3 (17) | 3 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Psychomotor skills impaired (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatillomania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/6 (0) | 0/3 (0) | 1/3 (1) | 0/2 (0) | 0/6 (0) | 0/1 (0) | 0/4 (0) | 0/4 (0) | 0/3 (0) | 0/5 (0) | 0/1 (0) | 0/2 (0)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulval disorder (Reproductive system and breast disorders) | 0/2 (0) | 0/2 (0) | 0/1 (0) | 0/3 (0) | 1/12 (1) | 0/2 (0) | 0/8 (0) | 0/4 (0) | 0/3 (0) | 0/5 (0) | 0/4 (0) | 0/8 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0/2 (0) | 0/2 (0) | 0/1 (0) | 0/3 (0) | 0/12 (0) | 0/2 (0) | 0/8 (0) | 0/4 (0) | 0/3 (0) | 0/5 (0) | 0/4 (0) | 1/8 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (5) | 4 (5) | 1 (6) | 2 (3) | 4 (4) | 0 (0) | 2 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (5) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (3) | 1 (3) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 3 (3) | 1 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (3) | 2 (2) | 1 (2) | 3 (6) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 4 (5) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (8) | 2 (3) | 1 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (4) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated without triggering the dose expansion cohorts for Parts D and E due to business considerations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review and comment on results communications prior to public release and can embargo communications regarding trial results for a period that is more than 30 days but less than or equal to 90 days from the time the sponsor receives the publication for review. The sponsor can request that the PI hold publishing the communication in order to protect any intellectual property interest at stake.

DOCUMENTS (2):
  • Study Protocol (2016-03-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT02784795/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT02784795/SAP_001.pdf